CLINICAL TRIAL: NCT05030532
Title: Expert Peer Facilitation of the EVERYbody Project: A Randomized-controlled Evaluation of a Diversity-focused, Dissonance-based, Universal Body Image Program for College Students
Brief Title: Expert Peer Facilitation of the EVERYbody Project
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In-person intervention activities halted in March 2020 due to COVID-19; follow-up data collection of active participants completed online in June 2020.
Sponsor: Western Washington University (Other)
Responsible Party: Principal Investigator, Anna Ciao, Associate Professor of Psychology, Western Washington University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-004_3
Record Dates: First submitted 2021-08-05; First posted 2021-09-01 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Body Image; Eating Disorder Symptom
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: After signing up for a specific time slot, participants were randomized in blocks of 20 to the EVERYbody Project or video comparison condition (two blocks of 10 participant slots were available in each time slot)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVERYbody Project: Expert facilitator version (Experimental): This gender inclusive, dissonance-based body image program was created from focus group feedback. Based on the Body Project, the program retains key dissonance activities while expanding the inclusivity focus (e.g., expanding the gender focus, exploring diversity within appearance ideals, critically discussing the impact of limited diversity representation in cultural appearance norms).
  Around 10% of content from the previous trial was modified to form the current intervention. Changes focused on enhancing diversity-focused content. College students with body image content interest completed two days (16 hours) of training on the program manual, group management, and conducting inclusive conversations. Post training, students self-assessed their facilitation readiness and were evaluated by two trainers on facilitation expertise. Peer leaders with sufficient expertise were invited to facilitate EVERYbody Project groups.
  Interventions: Behavioral: EVERYbody Project
- Video + Expressive Writing group (Active Comparator): Video + expressive writing groups were facilitated by a peer leader following a detailed script. This intervention was designed as an active but low-dissonance comparison condition. Participants viewed two separate documentary movies related to gender and/or appearance-related pressures (one during each session): (1) The Illusionists, and (2) The Mask You Live In. Participants engaged in a brief (10 minute) reflective writing exercise after each film. In order to keep dissonance low, participants were told that their reflections would not be shared with anyone and they were not turned in.
  Peer facilitators received brief (1 hour) training on the video group manual.
  Interventions: Other: Video + Expressive Writing

INTERVENTIONS:
Behavioral: EVERYbody Project — Brief behavioral group intervention (4 hours across two meetings)
  Arms: EVERYbody Project: Expert facilitator version
Other: Video + Expressive Writing — Brief video-based group intervention (4 hours across two meetings)
  Arms: Video + Expressive Writing group

SUMMARY:
The third trial of the EVERYbody Project explored the efficacy of using expert peer leaders to deliver the two-session, inclusive, group body image intervention compared to a time-matched video and expressive writing group through three-month follow-up. Expert peer leaders were college students with lived and/or academic expertise who were screened for facilitation readiness through a two-day training.

DETAILED DESCRIPTION:
The first two trials of the EVERYbody Project demonstrated that a gender-inclusive, diversity-focused, dissonance-based group body image intervention could improve eating disorder risk factors among college students, particularly when the two session program was delivered by individuals with expertise (faculty or staff with body image expertise). When peer interventionists were used (college students with body image interest who completed a two-day training before facilitating groups), the effects of the EVERYbody Project were diminished. Although peer facilitation is commonly used for delivering dissonance-based body image interventions, an open training peer facilitation model (where all students who are trained are eligible to deliver the intervention) may not be the most beneficial for leading inclusivity-focused body image groups.

The current trial of the EVERYbody Project (Trial 3) explores a novel strategy to implement this program using expert peer facilitators. College students with lived or academic expertise in both body image and diversity topics were recruited to complete a two-day training. The training included practice and feedback on the two session intervention content as well as training on inclusive facilitation. Following the training, peer leaders completed a facilitation readiness self-evaluation and were evaluated by trainers for facilitation expertise. Only students who passed the expertise threshold were invited to facilitate EVERYbody Project groups.

The expert peer facilitation of the EVERYbody Project was compared to a time-matched two session passive video and expressive writing intervention. College students within a university in the Pacific Northwest United States were invited to participate in the group intervention (universal intervention target, gender inclusive). Outcome assessment included a comparison of changes in eating disorder risk factors and symptoms across randomization conditions from pre-post intervention through three-month follow-up. Program satisfaction was assessed at post-intervention and program application was assessed post-intervention and at three-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Current college student enrolled at institution where research was taking place

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Eating disorder symptoms | Change from baseline through post-intervention (1-2 weeks) and follow-up (3 months)
  Eating disorder symptoms were assessed with an 8-item version of the Eating Disorders Examination Questionnaire (EDEQ). The 8-item version of the EDEQ yields a Global score (average across all 8 items).
Body Dissatisfaction | Change from baseline through post-intervention (1-2 weeks) and follow-up (3 months)
  The Satisfaction and Dissatisfaction with Body Parts Scale (SDBPS) assessed satisfaction and dissatisfaction with nine parts of the body that are commonly endorsed as concerning (e.g., stomach, thighs, hips). The average score was used in this study (average across all 9 items).
Internalized cultural appearance norms | Change from baseline through post-intervention (1-2 weeks) and follow-up (3 months)
  The two Internalization subscales of the Sociocultural Attitudes Toward Appearance Questionnaire-4 (SATAQ-4) assess internalized cultural messages surrounding appearance and attractiveness. The two internalization subscales were combined for this study (average across all 10 items), following prior research. This survey was assessed at all outcome time points (Survey 1, 2, and 3), plus midway through the intervention (following Session 1 of the program).
Negative affect | Change from baseline through post-intervention (1-2 weeks) and follow-up (3 months)
  Negative affect was assessed with 20 items from the fear, guilt, and sadness subscales of the Positive and Negative Affect Schedule-Revised (PANAS-X). The average of all 20 items was used in this study.

OTHER OUTCOMES:
Program satisfaction and application | Assessed at post-intervention (1-2 weeks after baseline) and follow-up (3 months)
  A series of feedback questions were used to gauge satisfaction with the EVERYbody Project after the second session (based on prior research). These questions included four Likert scale items about enjoyment (e.g., "I enjoyed the EVERYbody Project") rated from 1 (strongly disagree) to 5 (strongly agree) as well as open-ended questions (e.g., "Was any part of the EVERYbody Project particularly helpful/useful? If so, which part and why?") These questions were administered as a part of the post-intervention survey (Survey 2).
  At post-intervention (Survey 2) and three-month follow-up (Survey 3), three questions gauged application of information learned in the program (e.g., "How often do think about the things you learned in the EVERYbody Project?" rated on a scale from 1 (not at all) to 5 (all the time).

CONTACTS AND LOCATIONS:
Locations (1):
- Western Washington University, Bellingham, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and other materials will be made available following reasonable request to study Principal Investigator. All outcome data will be included in data sharing. Socio-demographic characteristics will be collapsed into broader categories to protect participant identity.
  Other study materials, including intervention manuals, will be housed on the Principal Investigator's Open Science Framework page, where URLs will be made publicly available.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Since the trial is complete, data are available immediately upon request.
URL: https://osf.io/x3k7v/?view_only=c9dbd31a4ad94a08b16421d719bc0fac

REFERENCES:
- [Background] Ciao AC, Munson BR, Pringle KD, Roberts SR, Lalgee IA, Lawley KA, Brewster J. Inclusive dissonance-based body image interventions for college students: Two randomized-controlled trials of the EVERYbody Project. J Consult Clin Psychol. 2021 Apr;89(4):301-315. doi: 10.1037/ccp0000636. PMID 34014692
- [Background] Ciao AC, Ohls OC, Pringle KD. Should body image programs be inclusive? A focus group study of college students. Int J Eat Disord. 2018 Jan;51(1):82-86. doi: 10.1002/eat.22794. Epub 2017 Nov 6. PMID 29105805
- [Background] Fairburn CG, Beglin SJ. Assessment of eating disorders: interview or self-report questionnaire? Int J Eat Disord. 1994 Dec;16(4):363-70. PMID 7866415
- [Background] Schaefer LM, Burke NL, Thompson JK, Dedrick RF, Heinberg LJ, Calogero RM, Bardone-Cone AM, Higgins MK, Frederick DA, Kelly M, Anderson DA, Schaumberg K, Nerini A, Stefanile C, Dittmar H, Clark E, Adams Z, Macwana S, Klump KL, Vercellone AC, Paxton SJ, Swami V. Development and validation of the Sociocultural Attitudes Towards Appearance Questionnaire-4 (SATAQ-4). Psychol Assess. 2015 Mar;27(1):54-67. doi: 10.1037/a0037917. Epub 2014 Oct 6. PMID 25285718
- [Background] Stice E, Shaw H, Burton E, Wade E. Dissonance and healthy weight eating disorder prevention programs: a randomized efficacy trial. J Consult Clin Psychol. 2006 Apr;74(2):263-75. doi: 10.1037/0022-006X.74.2.263. PMID 16649871
- [Background] Berscheid, E., Hatfield [Walster], E., & Bohrnstedt, G. (1973). The happy American body: A survey report. Psychology Today, 7, 119-131.
- [Background] Watson, D., & Clark, L. A. (1992). Affects separable and inseparable: On the hierarchical arrangement of the negative affects. Journal of Personality and Social Psychology, 62, 489-505. http://dx.doi.org/10.1037/ 0022-3514.62.3.489
- [Background] Kliem S, Schmidt R, Vogel M, Hiemisch A, Kiess W, Hilbert A. An 8-item short form of the Eating Disorder Examination-Questionnaire adapted for children (ChEDE-Q8). Int J Eat Disord. 2017 Jun;50(6):679-686. doi: 10.1002/eat.22658. Epub 2017 Jan 25. PMID 28122128
- [Background] Becker CB, Stice E. From efficacy to effectiveness to broad implementation: Evolution of the Body Project. J Consult Clin Psychol. 2017 Aug;85(8):767-782. doi: 10.1037/ccp0000204. PMID 28726480
- [Background] Kilpela LS, Blomquist K, Verzijl C, Wilfred S, Beyl R, Becker CB. The body project 4 all: A pilot randomized controlled trial of a mixed-gender dissonance-based body image program. Int J Eat Disord. 2016 Jun;49(6):591-602. doi: 10.1002/eat.22562. Epub 2016 May 18. PMID 27188688